CLINICAL TRIAL: NCT07047898
Title: The Effect of Dexmedetomidine on Postoperative Cognitive Function in Geriatric Patients Undergoing Robotic Urologic Surgery
Brief Title: The Effect of Dexmedetomidine on Postoperative Cognitive Function in Geriatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Muruvvet Taskir Turan, Principal investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-072
Record Dates: First submitted 2025-04-10; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Dexmedetomidine; Robotic Surgery; Geriatric Patients
Keywords: Postoperative Cognitive Function; recovery

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group receiving dexmedetomidine infusion (Active Comparator): Dexmedetomidine is a perioperative drug used for patients undergoing surgery under general anesthesia, which plays a role in brain and nerve protection. Dexmedetomidine is an α2-adrenergic agonist that pharmacologically exhibits effects such as sedation, analgesia, anxiolytic and diuresis, and has also been shown to have neuroprotective effects.
  Interventions: Drug: The group receiving dexmedetomidine infusion
- The group not receiving dexmedetomidine infusion (Active Comparator): Standard anesthesia maintenance will be applied
  Interventions: Drug: The group not receiving dexmedetomidine infusion

INTERVENTIONS:
Drug: The group receiving dexmedetomidine infusion — Dexmedetomidine will be administered intravenously at an infusion dose of 0.2-0.7 µg/kg/hour during the maintenance phase of anesthesia.
  Arms: The group receiving dexmedetomidine infusion
Drug: The group not receiving dexmedetomidine infusion — Infusion will not be given.
  Arms: The group not receiving dexmedetomidine infusion

SUMMARY:
In pelvic surgeries, using laparoscopic surgical procedures provides advantages such as reduced postoperative pain and complications, early mobilization, shorter hospital stays, lower costs, better cosmetic outcomes, and faster return to daily activities. In robotic surgeries, the instruments have superior maneuverability compared to the human wrist, allowing for more precise work in delicate areas with a three-dimensional view while eliminating the surgeon's hand tremor. On the other hand, despite advances in surgical techniques, anesthesia management, and intensive care, a significant proportion of geriatric patients experience cognitive decline after surgery. Postoperative cognitive function decline can reduce the quality of life and lead to significant damage to family and social support systems. Postoperative cognitive dysfunction (POCD), defined as a decline in cognitive function following surgeries performed under general anesthesia, is a common postoperative cognitive impairment, particularly in the elderly population. Studies have shown that the incidence of POCD in individuals aged 60 and above ranges between 20% and 40%. Additionally, POCD is associated with prolonged hospital stays, reduced mobility, and increased mortality. Patients undergoing robotic laparoscopic radical surgery assume the Trendelenburg position, which provides better exposure of the pelvic organs. However, in robotic-assisted laparoscopic surgeries, patients must be placed in a steep Trendelenburg position. Prolonged pneumoperitoneum and excessive head-down tilt can increase the permeability of the blood-brain barrier. As a result of the Trendelenburg position, intracranial pressure may increase, leading to brain hypoxia, inadequate cerebral blood flow, low arterial oxygen content, anemia, and high brain oxygen consumption. Impaired cerebral oxygenation can directly affect brain function. Compared to conventional laparoscopic surgery, patients undergoing robotic-assisted laparoscopic surgery tend to exhibit prolonged emergence from anesthesia and increased psychomotor agitation due to factors such as stress response, trauma, anesthesia, bleeding, and transfusion. This condition is influenced by factors such as decreased cerebral blood flow and hypotension. Therefore, real-time monitoring methods are needed to detect and address cerebral hypoxia. While diagnostic tools like computed tomography (CT), echocardiography (ECHO), electroencephalography (EEG), and magnetic resonance imaging (MRI) reveal brain damage at a later stage, near-infrared spectroscopy (NIRS) is a continuous, safe, and non-invasive method for detecting cerebral hypoxia. Identifying oxygen deficiency in the brain can allow adjustments in treatment strategies and help prevent postoperative cognitive dysfunction, potentially reducing patients' intensive care and hospital stay durations while minimizing complications. Recently, certain medications have been used to prevent postoperative cognitive dysfunction. Dexmedetomidine, a drug with neuroprotective properties, is commonly used perioperatively in patients undergoing surgery under general anesthesia. Pharmacologically, dexmedetomidine is an α2-adrenergic agonist with sedative, analgesic, anxiolytic, and diuretic effects. However, previous clinical studies evaluating the effects of dexmedetomidine on POCD in elderly patients have yielded inconsistent results. This study aims to investigate the effects of dexmedetomidine on recovery from anesthesia and postoperative cognitive function in elderly patients undergoing robotic urologic surgery, particularly focusing on its neuroprotective properties. Patients included in our study will be randomly divided into two groups. Both groups will undergo routine standard ASA monitoring, NIRS, and BIS monitoring. Both groups will receive standard anesthesia induction. Then, one group will receive sevoflurane + remifentanil, while the other group will receive dexmedetomidine and remifentanil infusion along with sevoflurane. Both patient groups will undergo the Mini-Mental State Examination (MMSE) before and after the operation. During the intraoperative period, anesthesia depth will be monitored using BIS (maintaining the depth between 40 and 60 for both groups), and oxygenation will be tracked using NIRS. Our study will include geriatric patients undergoing robotic urologic surgery. The patients will be randomly divided into two groups. The randomization process will be performed using a web-based randomization program (Sortition), which is defined for validity. The anesthesiologist providing anesthesia management and the anesthetist conducting the postoperative cognitive function monitoring will be different individuals. Patients who accept the study and undergo the preoperative Mini-Mental Test will be included in the study after postoperative assessments on the 24th hour and the 7th day.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years of age
* Those with ASA 1,2,3
* Patients who underwent robotic urological surgery
* Those who underwent Mini Mental Test in the preoperative period

Exclusion Criteria:

* Those under 65 years of age
* Those with ASA score IV and above
* Those with advanced co-morbidities
* Patients who have converted robotic surgery to open surgery
* Those with morbid obesity
* Those with alcohol or drug addiction
* Refusing to participate
* Those with a known history of psychiatric and neurological diseases
* Those with visual and hearing impairments
* Those who score below 24 on the Mini Mental Test
* Patients who are hemodynamically unstable peroperatively

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Postoperative cognitive dysfunction | preoperative 24 hour postoperative 24th hour and 7th day
  In order to evaluate cognitive impairment in patients who have undergone Mini Mental Test (0-30) in the preoperative 24 hour , the mini mental test will be performed again at the 24th hour and 7th day postoperatively.

SECONDARY OUTCOMES:
Recovery time | postoperative 30 minute
  The patient's recovery after extubation will be evaluated with the Ramsey sedation scale(1-6)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Yenimahalle, Ankara, Turkey (Türkiye)